CLINICAL TRIAL: NCT05015153
Title: Impact on Quality of Life with Pulmonary RehAbilitation After Pulmonary EMBOlism: RAMBO Study
Acronym: RAMBO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 29BRC21.0093 (RAMBO)
Record Dates: First submitted 2021-08-11; First posted 2021-08-20 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Embolism; Quality of Life and Dyspnea
MeSH Terms: conditions — Pulmonary Embolism; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): 20 sessions of Pulmonary rehabilitation will be performed over a period of 3 months
  Interventions: Other: Pulmonary rehabilitation (PR)
- Control group (No Intervention): No Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation (PR) — 20 sessions of PR in respiratory rehabilitation centre will be performed over a period of 3 months
  Arms: Intervention group

SUMMARY:
Pulmonary Embolism (PE) is a common and serious disease. Indeed, the annual incidence is 1/1000 patients per year and the 3-month mortality is 10%, which is twice that of myocardial infarction. The treatment is based on anticoagulation for at least 3 months. However, after three or six months of anticoagulation, persistent dyspnea and impairment of quality of life are observed in at least 30% of cases. Several mechanisms explain dyspnea and impairment of quality of life after PE, such as residual pulmonary artery obstruction, exercise deconditioning, depressive syndrome or development of a cardio-respiratory pathology. Pulmonary rehabilitation (PR) has been shown to be effective on dyspnea and quality of life and is included in the therapeutic management of chronic respiratory diseases such as Chronic Obstructive Pulmonary Disease (COPD) or pulmonary fibrosis. Furthermore, PR is also used after a myocardial infarction. However, PR after PE is still not included in therapeutic management of PE while outpatient management is recommended for the majority of patients after an acute PE episode. Study hypothesis is that PR has the potential to improve quality of life and dyspnea perception in patients who have received anticoagulation for at least 3 months after PE and who present an impairment of quality of life and/or a persistent dyspnea. This study presents several innovative aspects. First, to our knowledge, This study is the first large randomized trial assessing PR at least 3 months after acute symptomatic PE. Only one small randomized trial on 18 patients evaluating the impact of PR after PE has been published; as PR was performed just after the acute phase of PE in this trial, the clinical status improvement observed in this study could not be explained by PR alone, but also by anticoagulation. In this study, the investigators will include 112 patients at least 3 months after PE in order to exclude the bias related to anticoagulation effect. Second, This study is the first large randomized trial. Third, this study is the first that have the potential to demonstrate efficacy and safety of delayed PR after PE in patients with impaired quality of life due to persistent residual dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient treated with at least 3 months and up to 8 months of anticoagulation for symptomatic EP diagnosed according the ESC and ACCP guidelines.
* Patients who have a PembQol score ≥ 10% and whose total scores for the subgroups Q7+8 (dyspnea) and Q4 (impact of daily life) are ≥ 10%.

Exclusion Criteria:

* Presence of CTEPH according to international guidelines
* Patients treated for acute PE with anticoagulants for more than 8 months
* Active cancer or in remission for less than two years
* Dyspnea post - COVID due to parenchymal injuries
* Post-COVID hyperventilation syndrome without pulmonary vascular perfusion sequelae.
* Physical or psychological inability to undertake PR
* Isolated or more distal segmental PE
* Neuro-muscular disease with PR contraindication.
* Cardiac insufficiency (unstable coronary artery disease)
* Severe respiratory failure (long-term oxygen therapy, pulmonary hypertension)
* Chronic dyspnea MMRC ≥ 2 before PE
* Cardiac or respiratory rehabilitation in the previous year
* Indication to urgent PR within 6 months at the time of inclusion
* Life expectancy of less than 12 months
* Inability to give consent
* Patient under guardianship or curatorship
* Patient deprived of liberty by an administrative or judicial decision
* Patient has not social security affiliation or who don't beneficiary of such social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Quality of life - PEmbQoL score | 3 months
  Pulmonary embolism Quality of life score. This score includes 6 items regarding the frequency of lung complaints, their intensity, their physical, personal, social and professional impact. For each item, an average score is collected

SECONDARY OUTCOMES:
Safety : number and type of adverse reactions | 3 months
  Number of events
Quality of life - PEmbQoL score | 15 months
  Pulmonary embolism Quality of life score. This score includes 6 items regarding the frequency of lung complaints, their intensity, their physical, personal, social and professional impact. For each item, an average score is collected
Pulmonary Vascular Obstruction index | 3 months
  Pulmonary Vascular Obstruction (Meyer score) assessed with V/Q lung scan
Incidence of dyspnea | 3 months and 15 months
  Multidimensional dyspnea Profile (MDP) at the cycloergometer, Borg scale at the cycloergometer and at the 6 minute-walk-test, and Modified Medical Research Council scale (MMRC)
Change of 6 Minutes Walk Test | 3 months and 15 months
  6 Minutes Walk Test
Change of Psychological status | 3 months and 15 months
  Score of Hospital Anxiety and Depression scale. 14 rated items from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), allowing thus obtaining two scores (maximum score for each score = 21)
Symptomatic recurrent PE | 15 months
  Number of events
Arterial thromboembolic events | 15 months
  Number of events
Deaths of all causes | 15 months
  Number of events
Hospitalizations and acute medical events | 15 months
  Number of events

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Brest, Brest, France
  - CHU Angers, Angers
  - CHU de Grenoble, Grenoble
  - CHBS Lorient, Lorient
  - CH Morlaix, Morlaix
  - Hegp (Ap-Hp), Paris
  - Centre de santé de Roscoff, Roscoff
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.